CLINICAL TRIAL: NCT02087657
Title: Pilot Study Exploring the Use of Hyperbaric Oxygen in Autologous Peripheral Blood Stem Cell Transplant
Brief Title: Pilot Study Exploring the Use of Hyperbaric Oxygen in Autologous Peripheral Blood Stem Cell Transplantation
Acronym: Auto-HBO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Kansas Medical Center (Other)
Collaborators: SWOG Cancer Research Network (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Auto-HBO
Record Dates: First submitted 2014-03-12; First posted 2014-03-14 (Estimated); Last update posted 2017-02-14 (Actual); Status verified 2017-02

CONDITIONS: Multiple Myeloma; Hodgkin's Disease; Non-Hodgkin's Lymphoma
Keywords: Peripheral Blood Stem Cell (PBSC) Transplant; Hyperbaric oxygen; Lymphoma; Myeloma
MeSH Terms: conditions — Multiple Myeloma; Hodgkin Disease; Lymphoma, Non-Hodgkin; Lymphoma; Neoplasms, Plasma Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Hyperbaric Oxygen Treatment (Experimental): Administration of hyperbaric oxygen on the morning of stem cell transplant (Day 0).
  Interventions: Device: Administration of hyperbaric oxygen

INTERVENTIONS:
Device: Administration of hyperbaric oxygen — Hyperbaric oxygen at 2.5 atmospheres absolute (ATA) for a total of 2 hours
  Other Names: Monoplace Hyperbaric Chamber Model 3200 and 3200R

SUMMARY:
By doing this study, researchers hope to learn the following:

* The safety of hyperbaric oxygen administration in the setting of the autologous transplant
* The effects of hyperbaric oxygen administration on neutrophil count recovery and engraftment

DETAILED DESCRIPTION:
The post stem cell transplant complications of neutropenic fever and mucositis, related to the chemotherapy and/or radiation on hematopoietic tissue administered prior to peripheral blood stem cell transplant, are reversible upon neutrophil count recovery. The investigators will investigate the use of hyperbaric oxygen as an intervention to shorten neutropenia post-high-dose chemotherapy and autologous peripheral blood stem cell transplant. The idea of using hyperbaric oxygen therapy in autologous stem cell transplantation is based on the investigators pre-clinical work that supported the use of hyperbaric oxygen to improve umbilical cord blood (cluster of differentiation 34) CD34+ stem cell transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary written informed consent
* Subjects with Multiple Myeloma (MM), Hodgkin's Disease (HD), and non-Hodgkins lymphoma (NHL) who are eligible for high-dose chemotherapy and autologous PBSC transplant. Subjects should be enrolled within 30 days of transplant.
* Subjects must be >/= 18 yrs old and </= 70 yrs old
* Karnofsky performance status of >/= 70%
* Adequate hepatic, renal, cardiac and pulmonary function to be eligible for transplant. Minimum criteria include:

  * ALT (alanine aminotransferase), AST (aspartate aminotransferase): < 4x IULN (institutional upper limit of normal)
  * Total bilirubin: </= 2.0 mg/dL
  * Creatinine: </= 2.0 mg/dL
  * EF (ejection fraction) measured by 2D-ECHO or MUGA (multiple gated acquisition) scan of >/= 45%
  * FEV1 (forced expiratory volume), FVC (forced vital capacity) and DLCD(diffusing capacity of lung for carbon monoxide) >/= 50% of predicted value (corrected to serum hemoglobin)
* Women of child-bearing potential and men with partners of child-bearing potential must use adequate contraception prior to study entry and up to 30 days following treatment.

Exclusion Criteria:

* Pregnant or breast feeding
* Severe chronic obstructive pulmonary disease requiring oxygen supplementation
* History of spontaneous pneumothorax
* Active ear/sinus infection
* Claustrophobia
* HIstory of sinus or ear surgery, excluding myringotomy or ear tubes
* History of seizures

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-03; Primary Completion 2016-08 (Actual); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Presence or absence of a treatment limiting toxicity | Toxicity assessment occurs within 24hrs of treatment
  Treatment limiting toxicities are defined as the occurrence of any of the following complications within 24hrs of treatment: seizure disorder, pneumothorax, death, irreversible grade III or any grade IV toxicity that is determined by the treating physician to be at least likely related to HBO therapy.

SECONDARY OUTCOMES:
Reduction in time to neutrophil recovery and engraftment post-cord blood transplant. | Daily measurement of neutrophil counts, up to 40 days post transplant.
  Subjects will be followed daily until neutrophil recovery, defined as three consecutive days of achieving a neutrophil count of > 500/mm3. If subjects do not exhibit neutrophil recovery by Day 40 post transplant, they will be considered primary graft failures.

OTHER OUTCOMES:
Explore the effects of hyperbaric oxygen (HBO) therapy on erythropoietin (EPO) levels. | Assessment at: Day -7 (lymphoma) or Day -3 (myeloma), Pre-HBO (Day 0), Pre-transplant (6-10hrs post-HBO), 24 and 48 hrs after starting hyperbaric oxygen treatment as well as 3 days post-neutrophil engraftment
  Statistical methods will be applied to determine if the mean erythropoietin levels during the first 24 hours and 48 hours correlate with time to neutrophil recovery and engraftment.
Examine correlation between change to erythropoietin (EPO) levels and time to neutrophil recovery and engraftment. | EPO measurments: Pre-HBO (Day 0), 6-10hrs post-HBO, 24hrs and 48hrs post HBO, as well as 3 days post neutrophil engraftment.
  Erythropoietin blood levels will be correlated to the daily neutrophil counts to assess any relationship between erythropoietin levels and subsequent engraftment and neutrophil recovery.

CONTACTS AND LOCATIONS:
Overall Officials: Omar Aljitawi, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States